CLINICAL TRIAL: NCT00001170
Title: Affective Disorders and Affective Development: A Study of Child Rearing and Child Development in Normal Families and Families With Affective Disorders
Brief Title: Study of the Psychological Development of Children of Parents With and Without Affective Disorders
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 790123; 79-M-0123
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-02

CONDITIONS: Bipolar Disorder; Involutional Depression; Mood Disorder
Keywords: Parental Psychopathology; Child Rearing; Depression; Bipolar Affective Disorders; Manic-Depression; Social-Emotional Development; Cognitive Development; Child Psychopathology; Affective Disorder; Children at Risk
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Major; Mood Disorders; Depression

SUMMARY:
This research study is the continuation of a study started more than 20 years ago. The study was designed to explore the effect that depressed parents have on their children and to better understand the factors that contribute to depression development and maintenance.

The study will continue to investigate if children have certain characteristics in early and middle childhood that predict the later development of psychological disorders.

In addition, the study will continue looking at the processes responsible for the development of children of parents with and without affective (mood) disorders.

DETAILED DESCRIPTION:
The psychological development of offspring of parents with and without affective disorder is assessed from early childhood to young adulthood. Parents with a diagnosis of major depression or bipolar illness and well parents and their children are studied (SADS-L, RDC, and SCID, DSM-III). A sibling pair is studied in each family. Parent-child interaction is investigated through direct observation of behavior in naturalistic and controlled settings. Family history information is obtained through parent interviews. Behavioral observations, standard tests, physical examinations, and psychiatric interviews, and MRI procedures provide multiple assessments of the offspring. The study has been completed through preadolescence, adolescence, and late adolescence. Follow-up in young adulthood continues.

ELIGIBILITY:
Patients will be drawn from an ongoing longitudinal study begun in 1979 of offspring of parents with affective illness (unipolar and bipolar) and children of normal control parents.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1045
Dates: Start 1979-10; Study Completion 2005-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Achenbach TM, Edelbrock CS. The Child Behavior Profile: II. Boys aged 12-16 and girls aged 6-11 and 12-16. J Consult Clin Psychol. 1979 Apr;47(2):223-33. doi: 10.1037//0022-006x.47.2.223. No abstract available. PMID 469068
- [Background] Beardslee WR, Bemporad J, Keller MB, Klerman GL. Children of parents with major affective disorder: a review. Am J Psychiatry. 1983 Jul;140(7):825-32. doi: 10.1176/ajp.140.7.825. PMID 6344660
- [Background] Billings AG, Moos RH. Comparisons of children of depressed and nondepressed parents: a social-environmental perspective. J Abnorm Child Psychol. 1983 Dec;11(4):463-85. doi: 10.1007/BF00917076. PMID 6655148
- [Derived] Labella MH, Ruiz SK, Harris SJ, Klimes-Dougan B. Emotion socialization in mothers with mood disorders: Affective modeling and recollected responses to childhood emotion. Dev Psychopathol. 2021 Oct;33(4):1156-1169. doi: 10.1017/S0954579420000395. PMID 32672147
- [Derived] Klimes-Dougan B, Long JD, Lee CY, Ronsaville DS, Gold PW, Martinez PE. Continuity and cascade in offspring of bipolar parents: a longitudinal study of externalizing, internalizing, and thought problems. Dev Psychopathol. 2010 Nov;22(4):849-66. doi: 10.1017/S0954579410000507. PMID 20883586